

## **Informed Consent Form for Participants**

**Full Title of Project:** Evaluation of NAVIFY® Oncology Hub using simulation-based research methods

## Name of Principal Investigator:

Dr Saira Ghafur

Sponsor:

Prova Health Limited

Funder:

Roche/Genentech

**Initials** 

| 1. | I confirm that I have read and understand the participant information |
|---|---|
| | sheet dated 11 August 2022 version 2.0 for the above study and have |
| | had the opportunity to ask questions which have been answered fully. |
| 2. | l understand that my participation is voluntary, and l am free to |
| | withdraw at any time, without giving any reason and without my legal |
| | rights being affected. |
| 3. | l agree to take part in a simulated clinical scenario in which I will use |
| | NAVIFY® Oncology Hub |
| 4. | I agree to take part in a survey and brief interview to provide my |
| | feedback about the study as well as my thoughts about the NAVIFY® |
| | Oncology Hub application. |
| 5. | I understand I will receive financial compensation for taking part in this |
| | study. |
| 6. | I give consent for a screen recording of this session to be taken for the |
| | purposes of study analysis. |
| 7. | I understand that my participation is anonymous and any quotes from |
| | my survey or interview responses will be reported alongside my |
| | professional title only (e.g., Breast Oncologist, Major Cancer Center). |
| I | |

Version No: v2.0 Date: 11 August 2022



| Name of person taking consent | <br>Signature | <br>Date | |
|---|---|---|---|
| Name of interviewee | Signature | Date | |
| | | | _ |
| 0. I <b>give/do not give (OPTIONAL)</b> consent to being contacted to take part in other research studies conducted by Prova Health Limited | | | |
| purposes of informing produc | · | · | |
| shared with Roche/Genentech | | | |
| 9. give/do not give (OPTIONAL | L) consent for the sci | reen recording to be | |
| devices and stored securely at | Prova Health Limite | d. | |
| be kept confidential and store | d securely on passw | ord-protected | |
| 8. I understand that my personal | l data (i.e., name and | l email address) will | |

Version No: v2.0 Date: 11 August 2022